CLINICAL TRIAL: NCT02721420
Title: Malaria Chemoprevention With Monthly Treatment With Dihydroartemisinin-Piperaquine for the Post-discharge Management of Severe Anaemia in Children Less Than 5 Years in Malawi
Brief Title: Delivery of Malaria Chemoprevention in the Post-discharge Management of Children With Severe Anaemia in Malawi
Acronym: PMC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kamuzu University of Health Sciences (Other)
Collaborators: University of Bergen (Other); The Research Council of Norway (Other); Makerere University (Other); Liverpool School of Tropical Medicine (Other); Kenya Medical Research Institute (Other); University of Amsterdam (Other); Imperial College London (Other); London School of Hygiene and Tropical Medicine (Other); University of Minnesota (Other); Ministry of Health and Population, Malawi (Other Government); Ministry of Health, Malawi (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: P.02/15/1679
Record Dates: First submitted 2016-02-13; First posted 2016-03-29 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Malaria; Severe Anemia
MeSH Terms: conditions — Malaria; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Drug + short message(SMS) reminder (Other): dihydroartemesinin-piperaquine (3-day treatment courses, given 2, 6, and 10 weeks after enrolment) with SMS reminders prior to each treatment course
  Interventions: Drug: dihydroartemisinin-piperaquine; Other: short message(SMS) reminder
- Drug + no short message(SMS) reminder (Other): dihydroartemisinin-piperaquine (3-day treatment courses, given 2, 6, and 10 weeks after enrolment) without SMS reminders prior to each treatment course.
  Interventions: Drug: dihydroartemisinin-piperaquine
- Drug+ Health worker reminder (Other): dihydroartemisinin-piperaquine (3-day treatment courses, given 2, 6, and 10 weeks after enrolment) with Health surveillance assistants reminders prior to each treatment course.
  Interventions: Drug: dihydroartemisinin-piperaquine; Other: Health worker reminder
- Drug at hospital + SMS reminder (Other): dihydroartemisinin-piperaquine (3-day treatment courses, given 2, 6, and 10 weeks after enrolment) collected at the outpatient department without an SMS reminders prior to each treatment course.
  Interventions: Drug: dihydroartemisinin-piperaquine
- Drug at Hospital+no SMS reminder (Other): dihydroartemisinin-piperaquine (3-day treatment courses, given 2, 6, and 10 weeks after enrolment) collected at the outpatient department with a short message reminder prior to each treatment course
  Interventions: Drug: dihydroartemisinin-piperaquine; Other: message(SMS) reminder

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine
Other: message(SMS) reminder
  Arms: Drug at Hospital+no SMS reminder
Other: Health worker reminder — Health surveillance assistants reminders prior to each treatment course
  Arms: Drug+ Health worker reminder
Other: short message(SMS) reminder
  Arms: Drug + short message(SMS) reminder

SUMMARY:
Background and rationale: Children hospitalised with severe anaemia in Africa are at high risk of readmission or death within 6 months after discharge. No strategy specifically addresses this post-discharge period. In Malawi, 3 months of post-discharge malaria chemoprevention (PMC) with monthly 3-day treatment courses of artemether-lumefantrine (AL) in children with severe malarial anaemia prevented 31% of deaths and readmissions. The effect was in addition to the effect of insecticide-treated bednets. There is now need to design and evaluate effective delivery mechanism for PMC within the health system.

DETAILED DESCRIPTION:
Objectives: The primary objective of the trial is to determine the optimum PMC delivery mechanism by comparing community- versus health facility-based strategies in order to inform policy.

Study Type: This is a single-centre, matched, cluster randomized, 5-arm, factorial design trial comparing the uptake of PMC-DHP delivered through health facility or community-based approaches with or without SMS/HSA reminders.

Site: 90 villages in the catchment areas of Zomba Central hospital in southern Malawi

Study Population:

Inclusion criteria: convalescent children aged less than 5 years and weighing >5 kg admitted with severe anaemia (haemoglobin<5g/dL / Ht<15%); clinically stable, able to take or switch to oral medication; post-transfusion Hb >5g/dL.

Exclusion criteria: blood loss due to trauma, malignancy, known bleeding disorders or sickle cell trait, known hypersensitivity to study drug, known heart conditions, non-resident in study area, previous participation in study, known need at enrolment for prohibited medication and scheduled surgery during the course of the study. HIV infection and cotrimoxazole prophylaxis are not exclusion criteria

Study Interventions:

All children will receive Dihydroartemisinin-piperaquine (3-day treatment courses, given 2,6 and 10 weeks after discharge) either:

1. at discharge + SMS Reminder;
2. at discharge + No SMS Reminder;
3. at discharge + HSA Reminder;
4. at OPD + SMS Reminder; or
5. at OPD + No SMS Reminder

Outcome Measures:

Primary: 100% of PMC drugs uptake (defined as administration of all 3-day treatment courses, given 2, 6 and 10 weeks after discharge) assessed by unannounced spot checks.

Follow-up procedures: Children will be followed up for 15 weeks by passive case detection in 2 phases: Pre-PMC (2 weeks between hospital admission and 2 weeks post-discharge); PMC (2-14 weeks post-discharge)

Sample Size: A sample size of 75 children per arm (375 total children) allows for a detection of 25% increase in uptake from 50% to 75% with 10% loss to follow-up (power 90%, α=0.05).

Data Analysis: The % of children receiving IPTpd according to schedule will be compared by relative risks (95% CI), adjusted for prognostic factors at baseline using log binomial or Poisson regression with adjustment for cluster effects

ELIGIBILITY:
Inclusion Criteria:

1. Haemoglobin <5.0g/dl or PCV <15%, or requirement for blood transfusion for other clinical reasons on or during admission to the hospital
2. Age between 4 months (inclusive) and 59 months (inclusive)
3. Body weight >5kgs

Screening (in-hospital):

1. Fulfilled the pre-study screening eligibility criteria
2. Clinically stable, able to switch to oral medication
3. Subject completed blood transfusion(s) in accordance with routine hospital practice
4. Able to feed (for breastfed children) or eat (for older children)
5. Absence of known cardiac problems
6. Provision of informed consent by parent or guardian

Randomization (at discharge):

1. Fulfilled screening eligibility criteria
2. Still clinically stable, able to take oral medication, able to feed (for breastfed children) or eat (for older children) and able to sit unaided (for older children who were able to do so prior to hospitalization

Exclusion Criteria:

1. Recognised specific other cause of severe anaemia (e.g. trauma, haematological malignancy, known bleeding disorder)
2. Known sickle cell
3. Child will reside for more than 25% of the 3.5months study period (i.e. 3 weeks or more) outside of catchment area Enrolment in the study (t=0) at discharge
4. Previous enrolment in the present study
5. Known hypersensitivity to study drug
6. Sickle cell disease
7. Known need at the time of enrolment for concomitant prohibited medication during the 14 weeks PMC treatment period.
8. On-going or planned participation into another clinical trial involving on-going or scheduled treatment with medicinal products during the course of the study (3.5 months from enrolment)
9. Known need, or scheduled surgery during the course of the study (3.5 months)
10. Suspected non-compliance with the follow-up schedule
11. Known heart conditions, or family history of congenital prolongation of the QTc interval

Ages: 4 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 375 (Estimated)
Dates: Start 2016-03-24 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of those with 100 % uptake of PMC drugs during the 15 weeks of the study period. | 15 weeks
  100 % uptake is defined as administration of all study drugs and compliance to study visits during the course of 15 weeks.

SECONDARY OUTCOMES:
Proportion of those with 60% uptake of PMC drugs during the 15 weeks of the study period. | 15 weeks
  60 % uptake is defined as administration of 6 or more [but less than 9] of the daily dosages out of the total of 9 during the 15 week study period.
Proportion of those with 30 % uptake of PMC drugs during the 15 week trial period. | 15 weeks
  30 % PMC uptake is defined as administration of 3 or more [but less than 6] of the daily dosages out of the total of 9 during the 15 week trial period.
Proportion of those with <30% uptake of PMC drugs during the 15 week trial period. | 15 weeks
  <30 % PMC uptake is defined as administration of less than 3 of the daily dosages out of the total of 9 assessed during the 15 week trial period.

OTHER OUTCOMES:
All-causes of deaths and all-causes of hospital re-admissions during the 15 week trial period. | 15 weeks
  Assessment of all children who die or are hospitalised during the trial period
Assessment of the added costs of the interventions to the health system and the individual patients by conducting interviews during the 15 week trial period. | 15 weeks
Assessment of how the study interventions are acceptable by patients and health workers by conducting focus group discussions and using self administered questionnaires during the 15 week trial period. | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kamija Phiri, PhD, Principal Investigator — University of Malawi
Locations (1):
- College Of Medicine,Training and Research Unit Of Excellence,Zomba Central Hospital, Zomba, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nkosi-Gondwe T, Robberstad B, Mukaka M, Idro R, Opoka RO, Banda S, Kuhl MJ, O Ter Kuile F, Blomberg B, Phiri KS. Adherence to community versus facility-based delivery of monthly malaria chemoprevention with dihydroartemisinin-piperaquine for the post-discharge management of severe anemia in Malawian children: A cluster randomized trial. PLoS One. 2021 Sep 10;16(9):e0255769. doi: 10.1371/journal.pone.0255769. eCollection 2021. PMID 34506503
- [Derived] Nkosi-Gondwe T, Robberstad B, Blomberg B, Phiri KS, Lange S. Introducing post-discharge malaria chemoprevention (PMC) for management of severe anemia in Malawian children: a qualitative study of community health workers' perceptions and motivation. BMC Health Serv Res. 2018 Dec 19;18(1):984. doi: 10.1186/s12913-018-3791-5. PMID 30567567
- [Derived] Gondwe T, Robberstad B, Mukaka M, Lange S, Blomberg B, Phiri K. Delivery strategies for malaria chemoprevention with monthly dihydroartemisinin-piperaquine for the post-discharge management of severe anaemia in children aged less than 5 years old in Malawi: a protocol for a cluster randomized trial. BMC Pediatr. 2018 Jul 20;18(1):238. doi: 10.1186/s12887-018-1199-3. PMID 30029620
- [Derived] Svege S, Kaunda B, Robberstad B, Nkosi-Gondwe T, Phiri KS, Lange S. Post-discharge malaria chemoprevention (PMC) in Malawi: caregivers; acceptance and preferences with regard to delivery methods. BMC Health Serv Res. 2018 Jul 11;18(1):544. doi: 10.1186/s12913-018-3327-z. PMID 29996833